CLINICAL TRIAL: NCT03173950
Title: Phase II Trial of the Immune Checkpoint Inhibitor Nivolumab in Patients With Recurrent Select Rare CNS Cancers
Brief Title: Immune Checkpoint Inhibitor Nivolumab in People With Recurrent Select Rare CNS Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170102; 17-C-0102
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06-26

CONDITIONS: Medulloblastoma; Ependymoma; Pineal Region Tumors; Choroid Plexus Tumors; Atypical/Malignant Meningioma
Keywords: Immunotherapy; Anti-PD-1 Antibody; Brain Tumors; MDASI-BT; Spinal Cord Tumors
MeSH Terms: conditions — Medulloblastoma; Ependymoma; Pinealoma; Choroid Plexus Neoplasms; Meningioma; Brain Neoplasms; Spinal Cord Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Experimental Therapy (Experimental): Individuals will receive nivolumab at standard dose of 240 mg IV every 2 weeks for cycles 1 through 2, then doses of 480 mg every 4 weeks for a total of 14 additional doses
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Individuals will receive nivolumab at standard dose of 240 mg IV every 2 weeks for cycles 1 through 2, then doses of 480 mg every 4 weeks for a total of 14 additional doses

SUMMARY:
Background:

More than 130 primary tumors of the central nervous system (CNS) have been identified. Most affect less than 1,000 people in the United States each year. Because these tumors are so rare, there are few proven therapies. This study will test whether the immunotherapy drug nivolumab is an effective treatment for people with rare CNS tumors.

Objectives:

To learn if stimulating the immune system using the drug nivolumab can shrink tumors in people with rare CNS (brain or spine) tumors or increase the time it takes for these tumors to grow or spread.

Eligibility:

Adults whose rare CNS tumor has returned.

Design:

Individuals will be screened:

* Heart and blood tests
* Physical and neurological exam
* Hepatitis tests
* Pregnancy test
* MRI. They will lay in a machine that takes pictures.
* Tumor tissue sample. This can be from a previous procedure.

At the start of the study, participants will have blood tests. They will answer questions about their symptoms and their quality of life.

Individuals will get nivolumab in a vein every 2 weeks for up to 64 weeks.

Individuals will have monthly blood tests. Every other month they will have an MRI and a neurologic function test. They will also answer questions about their quality of life.

Genetic tests will be done on individuals' tumor tissue. Individuals will be contacted if any clinically important results are found.

After treatment ends, individuals will be monitored for up to 5 years. They will have a series of MRIs and neurological function tests. They will be asked to report any symptoms they experience....

DETAILED DESCRIPTION:
Background:

* There are more than 130 identified primary tumors of the central nervous system (CNS). Most have an annual incidence of less than 1000 in the United States.
* Given the rarity of each of the tumors listed above, there is a paucity of proven therapies. Most of these neoplasms are treated with maximum surgical resection followed by treatment with external beam radiotherapy. With few exceptions (medulloblastoma, adult ependymoma), there are no effective systemic regimens and even in chemotherapy sensitive disease, most patients with recurrence eventually have no remaining salvage treatments available.
* In the setting of this unmet need, we propose to create a basket protocol that will evaluate the efficacy of the PD-1 inhibitor, nivolumab, in patients with refractory rare central nervous system neoplasms.
* This study seeks to establish effective therapies at recurrence in patients with rare CNS tumors. We hypothesize that this therapy will improve progression free survival and/or objective responses.
* It will be important to determine whether any determined survival benefit is associated with improvements in symptoms or does a worsening of symptoms offset the increase in survival. Precedence exists for measuring non-therapeutic endpoints in oncology research, and specifically in studies evaluating therapeutic benefit in patients with CNS tumors. There have been efforts in neuro-oncology to evaluate secondary endpoints using validated instruments as an additional indicator of benefit. The M.D. Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) and Spine Tumor Module (MDASI-SP) allow for the self-reporting of symptom severity and interference with daily activities for patients with either brain or spinal cord tumors. The availability of validated instruments provides an opportunity to prospectively assess the impact of treatment, both positive and negative, on patients.

Objective:

Determine the efficacy of nivolumab in a variety of recurrent, refractory primary central nervous system tumors as measured by disease control rate (confirmed CR/PR or durable SD for at least 6 months).

Eligibility:

* Documented recurrent or progressive disease that corresponds to one of the tumors eligible for testing.
* Age >= 18 years of age.
* Karnofsky Performance >= 70%.
* Tumor tissue available for central review to confirm morphologic diagnosis
* Tumor tissue or slides must be available for central molecular and immune profiling.

Design:

* This is an open label phase II clinical trial. Patients will be treated with the immune checkpoint inhibitor, nivolumab, at a standard dose of 240 mg intravenously every 2 weeks (+/- 3 days) for cycles 1 through 2, then doses of 480 mg every 4 weeks (+/- 3 days) for a total of 14 additional doses (cycles). A maximum of 18 treatments will be given (64 weeks).
* A cycle will be defined as 4 weeks and patients will undergo efficacy assessments using MR imaging (and/or other imaging tests if applicable) every 2 cycles. Toxicity assessments will occur before the initiation of each cycle and patient outcomes measures (PROs) will be completed at the time of each imaging study (every 2 cycles) but prior to the patient being informed of the imaging results.
* After completion of the planned treatment course or if treatment was stopped because of toxicity, patients will undergo imaging evaluations and PRO measurements every 8 weeks (or 2 months) for one year, then every 3 months for the next year, then every 4

months for the next year and then every 6 months while the patient remains on the protocol. Patients off treatment because of disease progression will not undergo future imaging or PRO assessments on this protocol.

* Bayesian Optimal Phase 2 design (BOP2), will be used to conduct this phase II trial in patients with a variety of recurrent, refractory primary central nervous system tumors.
* The study will be comprised of 2 disease cohorts: heavily pretreated (defined as having received 3 or more prior therapies) and non-heavily pretreated (defined as having received up to 2 prior therapies). Each cohort will be evaluated independently for efficacy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histopathologically proven diagnosis of Ependymoma, Medulloblastoma, Parenchymal Pineal Region Tumors (Pineoblastoma, Pineocytoma, Pineal Tumor of Intermediate Differentiation, Papillary Tumor of the Pineal Region), Choroid Plexus Tumors (Carcinoma, Papilloma, Atypical Papilloma), Histone Mutated Gliomas, Gliomatosis Cerebri, ATRT, Malignant/Atypical Meningioma*, Gliosarcoma or Primary CNS Sarcoma, Pleomorphic Xanthoastrocytoma (PXA) and Anaplastic Pleomorphic Xanthoastrocytoma (APXA), and tumors formerly known as Primitive Neuro-Ectodermal Tumors (Embryonal Tumor with Multilayered Rosettes, Medulloepithelioma, CNS Neuroblastoma, CNS Ganglioneuroblastoma, CNS Embryonal Tumor NOS; and tumor entities emerging from methylation profiling of CNS-PNETs: CNS neuroblastoma with FOXR2 activation, CNS Ewing sarcoma family tumor with CIC alteration, CNS high-grade neuroepithelial tumor with MN1 alterations, and CNS high-grade neuroepithelial tumor with BCOR alteration) prior to registration.

  *Individuals with extra CNS metastases from meningioma will be eligible even if pathology review fails to demonstrate high grade features on available tumor samples.
* The tumor tissue (e.g., block or 20 unstained slides) must be available to be sent for immunophenotyping by NCI Laboratory of Pathology.
* Individuals must have progressive tumor growth after having received established standard of care and/or other experimental treatments for their newly diagnosed or recurrent disease. Individuals will be enrolled into 2 different cohorts (cohort 1 or heavily pretreated; cohort 2 or not heavily pretreated).
* Age >= 18
* Karnofsky performance status >= 70 within 14 days prior to Step 2 registration; Individuals with severe paraparesis/paraplegia who need minimal assistance for selfcare due to their motor deficit but are otherwise functionally independent will be considered eligible.
* Adequate hematologic function based on CBC/differential within 14 days prior to Step 2 registration defined as follows:

  * Absolute neutrophil count >= 1,500 cells/mm3;
  * Platelet count >= 100,000 cells/mm3
  * Hemoglobin > 9.0 g/dl (may be transfused to achieve this level)
* Adequate renal function within 14 days prior to Step 2 registration defined as follows:

  * BUN <= 30 mg/dl and
  * Serum creatinine <= 1.7 mg/dl

Note: If the serum creatinine is greater than 1.7 mg/dl, a 24-hour urine creatinine clearance will be obtained and if the result of this study is within normal limits*, the patient would be eligible to enroll onto study. (*Normal Creatinine Clearance Range: Male: 90 - 130 ml/min; Female: 80 - 125 ml/min)

* Adequate hepatic function within 14 days prior to Step 2 registration defined as follows:

  * Total bilirubin (except patients with Gilbert's Syndrome, who are eligible for the study but exempt from the total bilirubin eligibility criterion) <= 2.0 mg/dl and
  * ALT and AST <= 2.5x ULN
* No active or chronic hepatitis infection. HCV antibody (for Hepatitis C) and Hepatitis B Surface antigen and Hepatitis B core antibody must be negative. This has been routinely incorporated into immunotherapy trials with checkpoint inhibitors because of concerns that the risk of treatment-induced hepatic injury is increased in the setting of active viral hepatitis.
* The individual must not be on a corticosteroid dose greater than physiologic replacement dosing defined as 30 mg of cortisone per day or its equivalent.
* The individual must provide study-specific informed consent prior to study entry. No Durable Power of Attorney or Next of Kin can provide initial consent.
* The effects of nivolumab on the developing human fetus are unknown. For this reason, women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 5 months (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug.

NOTE: Based on the evidence cited in Nivolumab IB ver. 20, given that nivolumab is not a genotoxic agent, and that relevant systemic concentrations sufficient to produce a risk of fetal toxicity are not expected in IOCBP partners from exposure to an individual's seminal fluid, men that can father children will not be required to use contraceptive measures and/or a latex or other synthetic condom during sexual activity with an WOCBP partner.

EXCLUSION CRITERIA:

* Individuals who are receiving any other investigational agents.
* Prior use of an immunotherapy such as (but not limited to) a vaccine therapy, dendritic cell vaccine, other checkpoint inhibitors, or intracavitary or convectional enhanced delivery of chemotherapy.
* Prior or concurrent malignancy unless its natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen.
* Severe, active co-morbidity defined as follows:

  * Unstable angina within the last 6 months prior to Step 2 registration.
  * Transmural myocardial infarction within the last 6 months prior to Step 2 registration.
  * Evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of >= 2 mm using the analysis of an EKG performed within 14 days prior to Step 2 registration.
  * New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to Step 2 registration.
  * History of stroke, cerebral vascular accident (CVA) or transient ischemic attack within 6 months prior to Step 2 registration, with the exception of pericavitary ischemia due to tumor resection.
  * Serious and inadequately controlled cardiac arrhythmia.
  * Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease.
  * Evidence of bleeding diathesis or coagulopathy.
  * Serious or non-healing wound, ulcer, or bone fracture or history of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Step 2 registration, with the exception of the craniotomy for tumor resection.
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration.
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects.
  * Known acquired immune deficiency syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude participants with AIDS is based on the lack of information regarding the safety of nivolumab in patients with active HIV infection.
  * Active connective tissue disorders, such as lupus or scleroderma, which in the opinion of the treating physician may put the patient at high risk for immunologic toxicity.
* Individuals with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to individuals with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome or CIDP, myasthenia gravis; systemic autoimmune disease such as SLE, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and individuals with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease.

Of note, individuals with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Participants with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible. However, individuals with vitiligo, diabetes mellitus, and Hashimoto thyroiditis on appropriate replacement therapy may be enrolled.

* Any other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy.
* Allergies and Adverse Drug Reaction: History of allergy to study drug components.
* Pregnancy or lactating women due to possible adverse effects on the developing fetus or infant due to study drug. Women of childbearing potential must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to Step 2 registration.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Individuals unable to have MRIs.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
objective response | end of treatment
  Rate of achieving a confirmed Complete Response/Partial Response (confirmed by imaging one month later)
progression free survival rate | 6 months after end of treatment
  Rate of durable Stable Disease lasting at least 6 months (PFS-6)

CONTACTS AND LOCATIONS:
Overall Officials: Byram H Ozer, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - UT MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Gilbert MR, Ruda R, Soffietti R. Ependymomas in adults. Curr Neurol Neurosci Rep. 2010 May;10(3):240-7. doi: 10.1007/s11910-010-0109-3. PMID 20425040
- [Background] Okada H, Weller M, Huang R, Finocchiaro G, Gilbert MR, Wick W, Ellingson BM, Hashimoto N, Pollack IF, Brandes AA, Franceschi E, Herold-Mende C, Nayak L, Panigrahy A, Pope WB, Prins R, Sampson JH, Wen PY, Reardon DA. Immunotherapy response assessment in neuro-oncology: a report of the RANO working group. Lancet Oncol. 2015 Nov;16(15):e534-e542. doi: 10.1016/S1470-2045(15)00088-1. PMID 26545842
- [Background] Daud AI, Loo K, Pauli ML, Sanchez-Rodriguez R, Sandoval PM, Taravati K, Tsai K, Nosrati A, Nardo L, Alvarado MD, Algazi AP, Pampaloni MH, Lobach IV, Hwang J, Pierce RH, Gratz IK, Krummel MF, Rosenblum MD. Tumor immune profiling predicts response to anti-PD-1 therapy in human melanoma. J Clin Invest. 2016 Sep 1;126(9):3447-52. doi: 10.1172/JCI87324. Epub 2016 Aug 15. PMID 27525433
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0102.html